CLINICAL TRIAL: NCT07067151
Title: Use of Noninvasive Wearables Biomonitoring to Detect Pre-Smoking, Smoking, And Post-Smoking Stages: An Observational Laboratory Study
Brief Title: Using Smartwatches to Monitor Smoking in Real-life Situations
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002323; 002323-MD
Record Dates: First submitted 2025-07-12; First posted 2025-07-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-26

CONDITIONS: Smoking
Keywords: Nicotine; Smoking; Smart watches; Pre-smoking; Cessation support; Thermal-sensor wearables; Home-based assessment; Cigarettes; Observational
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smokers: Individuals aged 21 and older who smoke, have not gone beyond a high school education, and earn low incomes.

SUMMARY:
Background: It is important to quickly identify when people are at risk of smoking. Most current methods rely on people reporting when they smoke or what makes them want to smoke. But this can be hard for people to do and may not always be accurate. Other methods use special gadgets to identify smoking movements, but these may not always work well in real life. We want to see if we can use devices available on the market such as smartwatches to identify signs in the body and hand movements that might indicate when someone is about to smoke, is currently smoking, or has just smoked.

Objective: To record body signs and hand movements before, during, and after smoking in real-life and in a lab to see how they change when someone is craving cigarettes, while a person is smoking, and after a person has smoked.

Eligibility: People who are 21 years or older and smoke, do not have more than a high school education, and are low-income earners. To participate in the study, participants have to pass a breath test that shows they smoke cigarettes and, for women, a urine test to show that they are not currently pregnant.

Design: Participants will complete an eligibility survey to see if they qualify to be in the study. If they qualify, they will answer a brief baseline survey that includes questions about themselves, their health, and their smoking behavior.

Participants will get a smartwatch to wear for 3 days at home, log each time they are about to smoke and have finished smoking, and answer a 5-question health survey via the app. They will get instructions on how to set up and wear the smartwatch. They will download a mobile application on their phone. The app will collect data from the smartwatch.

Participants will then come to the lab but will be asked not to smoke or drink alcohol for at least 12 hours. They will have to take a breath test to show they have not smoked or had alcohol. They will also give a blood sample. In the lab, they will sit in a room where they will be hooked to devices that monitor their vitals such as heart rate and blood pressure for one hour. They will also wear a smartwatch on each hand. While they are in the smoking room, they will go through 3 different phases: (a) pre-smoking where they will be asked to stay seated for about 25 minutes, (b) smoking where they will be asked to smoke as many cigarettes of their choice as they want for about 10 to 15 minutes, (c) post-smoking where they will be asked to stay seated, not smoking, for about 25 minutes. They will answer a brief 10-minute health survey before and after the session.

Participation will last for 3 days of home monitoring and 2 visits to the research clinic that last about 2 hours.

DETAILED DESCRIPTION:
Background:

The study is part of a systematic effort to develop and evaluate a smoking cessation intervention, Quit Journey, a smoking cessation intervention targeting individuals with low socioeconomic status. Specifically, the study will inform the development of just-in-time momentary support to preempt a lapse or prevent it from progressing to a relapse to users of Quit Journey. Additionally, the study fills a gap in wearable-based studies for smoking detection that have thus far relied exclusively on socially and economically advantaged populations by increasing the representation of underserved populations and more accurately developing algorithms for smoking detection that include input from minority populations and pave the way for its replication with a larger sample in real-world settings. Finally, the data collected from this laboratory-based study will serve as baseline parameters for detecting smoking events in free-living conditions. In a planned real-world study, we aim to finetune our smoking-detection algorithms with data collected in natural environments, potentially improving their robustness and generalizability. Insights from this study have real-world applications of smoking-detection algorithms in wearables and mobile applications, ultimately advancing technology-assisted smoking cessation and contributing to reduced smoking rates.

Objectives:

* The objective of this study is to identify wearables-based digital biomarkers that are associated with nicotine deprivation (i.e., pre-smoking) and satiation (i.e., post-smoking) and with smoking episodes (i.e., during smoking). Identifying signature digital biomarkers of smoking can help us to unobtrusively detect with great probability the proclivity to smoke or smoking behavior, which can inform the delivery of momentary support to preempt lapsing or progressing toward a relapse among people attempting to quit smoking.
* We hypothesize that, relative to pre-smoking, (a) blood oxygen saturation will be lower, (b) heart rate will be higher, (c) heart rate variability will be higher, and (d) respiratory rate will be lower during a smoking episode and post-smoking.

Endpoints:

* Primary endpoint: Changes in wearables-measured biomarker measures including heart rate, heart rate variability, respiratory rate, and blood oxygenation, in addition to hand/arm movement, across three smoking stages.
* Secondary endpoint: Not applicable.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will recruit up to 30 non-treatment seeking participants with low socioeconomic status who smoke. We will strive to have representation across racial and ethnic groups and biological sex.

To be included in the study, participants must:

* be 21 years or older in compliance with Tobacco 21 laws
* be maximally high school educated (or equivalent) and earn at or below 200% of the federal poverty line for 2024 corresponding to number of people in their household (US Department of Health and Human Services)
* have smoked 100 cigarettes in their lifetime and 5+ cigarettes per day in the past year to establish daily smoking status
* willing to abstain from smoking for >=12 hours prior to the lab visit verifiable by a CO reading that is below 10 ppm and retrospectively by minimal nicotine in blood sample
* willing to abstain from using any nicotine products or devices for (Bullet)12 hours prior to the lab visit
* willing to abstain from alcohol use for >=12 hours prior to the lab session verifiable by breath alcohol concentration (BrAC = 0.000)
* willing to adhere to all study procedures including agreeing to a blood draw and bringing >=1cigarette for use during the study visit
* have a smartphone compatible with wearable device requirements for Bluetooth and operating system (iphone iOS 14 and higher, Android 9.0 and higher) and willing to download the study apps onto their phone
* speak English
* and willing and able to provide informed consent.

Participants will be excluded if they:

* are not abstinent before the lab session through biochemical verification after two attempts
* have sought treatment for tobacco/nicotine use in the past 2 months (e.g., on pharmacotherapy for smoking cessation, enrolled in smoking cessation support programs or interventions, currently attempting to change their nicotine/tobacco use) or intend to quit within the next month
* have past 3-month pulmonary or cardiovascular event, or those who have been hospitalized or visited the emergency room for seizure, stroke, or new heart problems,
* are pregnant or breastfeeding
* and are unable or unwilling to provide informed consent.

EXCLUSION CRITERIA:

Vulnerable populations will not be enrolled in the study (i.e., adults unable to consent, individuals who are not yet adults, pregnant women, prisoners).

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise individuals aged 21 years or older who currently smoke cigarettes. Participants must have completed a high school education or possess a lower level of academic achievement, and they should be classified as low-income earners. To be eligible for participation in the study, individuals will need to successfully pass a breath test that confirms their smoking status. Furthermore, female participants will be required to undergo a urine test to verify that they are not currently pregnant, ensuring the study's safety and ethical standards. This rigorous participant selection process is designed to ensure a focused and relevant study group that aligns with the research objectives.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to evaluate changes in biomarker measurements obtained from wearables, which include heart rate, heart rate variability, respiratory rate, blood oxygen levels & hand/arm movement, across three smoking stages. | 7 days
  As the research progresses, the team will work diligently to gather a robust dataset from various sources, including wearable devices, lab sessions, medical-grade information, and detailed questionnaires. This comprehensive approach will enable the identification of specific biomarkers and hand-mouth gestures related to the different stages of tobacco use: pre-smoking, active smoking, and post-smoking. By analyzing these diverse data sources, the team aims to gain valuable insights into the physiological and behavioral patterns associated with each stage. This knowledge will not only enrich our understanding of tobacco use but also pave the way for developing targeted interventions and tailored support systems for individuals seeking to quit smoking. Through collaboration and innovative analysis, this research endeavors to create more effective strategies for smoking cessation, ultimately fostering healthier lifestyles.

CONTACTS AND LOCATIONS:
Overall Officials: Sherine M El-Toukhy, Ph.D., Principal Investigator — National Institute on Minority Health and Health Disparities (NIMHD)
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hojjatinia S, Daly ER, Hnat T, Hossain SM, Kumar S, Lagoa CM, Nahum-Shani I, Samiei SA, Spring B, Conroy DE. Dynamic models of stress-smoking responses based on high-frequency sensor data. NPJ Digit Med. 2021 Nov 23;4(1):162. doi: 10.1038/s41746-021-00532-2. PMID 34815538
- [Background] Hoeppner BB, Hoeppner SS, Seaboyer L, Schick MR, Wu GW, Bergman BG, Kelly JF. How Smart are Smartphone Apps for Smoking Cessation? A Content Analysis. Nicotine Tob Res. 2016 May;18(5):1025-31. doi: 10.1093/ntr/ntv117. Epub 2015 Jun 4. PMID 26045249
- [Background] Hoeppner BB, Hoeppner SS, Schick MR, Milligan CM, Helmuth E, Bergman BG, Abroms LC, Kelly JF. Using the text-messaging program SmokefreeTXT to support smoking cessation for nondaily smokers. Subst Use Misuse. 2019;54(8):1260-1271. doi: 10.1080/10826084.2018.1552300. Epub 2019 Apr 19. PMID 30999794
- [Background] Ho BK, Robinson JK. Color bar tool for skin type self-identification: A cross-sectional study. J Am Acad Dermatol. 2015 Aug;73(2):312-3.e1. doi: 10.1016/j.jaad.2015.05.024. No abstract available. PMID 26183973
- [Background] Henrich J, Heine SJ, Norenzayan A. Most people are not WEIRD. Nature. 2010 Jul 1;466(7302):29. doi: 10.1038/466029a. No abstract available. PMID 20595995
- [Background] Hebert ET, Stevens EM, Frank SG, Kendzor DE, Wetter DW, Zvolensky MJ, Buckner JD, Businelle MS. An ecological momentary intervention for smoking cessation: The associations of just-in-time, tailored messages with lapse risk factors. Addict Behav. 2018 Mar;78:30-35. doi: 10.1016/j.addbeh.2017.10.026. Epub 2017 Oct 28. PMID 29121530
- [Background] Hebert ET, Ra CK, Alexander AC, Helt A, Moisiuc R, Kendzor DE, Vidrine DJ, Funk-Lawler RK, Businelle MS. A Mobile Just-in-Time Adaptive Intervention for Smoking Cessation: Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Mar 9;22(3):e16907. doi: 10.2196/16907. PMID 32149716
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Hayano J, Yamada M, Sakakibara Y, Fujinami T, Yokoyama K, Watanabe Y, Takata K. Short- and long-term effects of cigarette smoking on heart rate variability. Am J Cardiol. 1990 Jan 1;65(1):84-8. doi: 10.1016/0002-9149(90)90030-5. PMID 2294686
- [Background] Grimes LM, Garg R, Weng O, Wolff JM, McQueen A, Carpenter KM, Kreuter MW. Appeal of Tobacco Quitline Services Among Low-Income Smokers. Prev Chronic Dis. 2023 Mar 2;20:E11. doi: 10.5888/pcd20.220214. PMID 36862604
- [Background] Galobardes B, Shaw M, Lawlor DA, Lynch JW, Davey Smith G. Indicators of socioeconomic position (part 1). J Epidemiol Community Health. 2006 Jan;60(1):7-12. doi: 10.1136/jech.2004.023531. PMID 16361448
- [Background] El-Toukhy S, Pike JR, Zuckerman G, Hegeman P. Decision Trade-Offs in Ecological Momentary Assessments and Digital Wearables Uptake: Protocol for a Discrete Choice Experiment. JMIR Res Protoc. 2023 Sep 25;12:e47567. doi: 10.2196/47567. PMID 37747771
- [Background] Dinas PC, Koutedakis Y, Flouris AD. Effects of active and passive tobacco cigarette smoking on heart rate variability. Int J Cardiol. 2013 Feb 20;163(2):109-15. doi: 10.1016/j.ijcard.2011.10.140. Epub 2011 Nov 17. PMID 22100604
- [Background] Cornelius ME, Loretan CG, Jamal A, Davis Lynn BC, Mayer M, Alcantara IC, Neff L. Tobacco Product Use Among Adults - United States, 2021. MMWR Morb Mortal Wkly Rep. 2023 May 5;72(18):475-483. doi: 10.15585/mmwr.mm7218a1. PMID 37141154
- [Background] Collins LM, Baker TB, Mermelstein RJ, Piper ME, Jorenby DE, Smith SS, Christiansen BA, Schlam TR, Cook JW, Fiore MC. The multiphase optimization strategy for engineering effective tobacco use interventions. Ann Behav Med. 2011 Apr;41(2):208-26. doi: 10.1007/s12160-010-9253-x. PMID 21132416
- [Background] Cole CA, Powers S, Tomko RL, Froeliger B, Valafar H. Quantification of Smoking Characteristics Using Smartwatch Technology: Pilot Feasibility Study of New Technology. JMIR Form Res. 2021 Feb 5;5(2):e20464. doi: 10.2196/20464. PMID 33544083
- [Background] Cole CA, Anshari D, Lambert V, Thrasher JF, Valafar H. Detecting Smoking Events Using Accelerometer Data Collected Via Smartwatch Technology: Validation Study. JMIR Mhealth Uhealth. 2017 Dec 13;5(12):e189. doi: 10.2196/mhealth.9035. PMID 29237580
- [Background] Cerrada CJ, Dzubur E, Blackman KCA, Mays V, Shoptaw S, Huh J. Development of a Just-in-Time Adaptive Intervention for Smoking Cessation Among Korean American Emerging Adults. Int J Behav Med. 2017 Oct;24(5):665-672. doi: 10.1007/s12529-016-9628-x. PMID 28070868
- [Background] Carter BL, Lam CY, Robinson JD, Paris MM, Waters AJ, Wetter DW, Cinciripini PM. Real-time craving and mood assessments before and after smoking. Nicotine Tob Res. 2008 Jul;10(7):1165-9. doi: 10.1080/14622200802163084. PMID 18629726
- [Background] Carreiro S, Fang H, Zhang J, Wittbold K, Weng S, Mullins R, Smelson D, Boyer EW. iMStrong: Deployment of a Biosensor System to Detect Cocaine Use. J Med Syst. 2015 Dec;39(12):186. doi: 10.1007/s10916-015-0337-9. Epub 2015 Oct 21. PMID 26490144
- [Background] Businelle MS, Perski O, Hebert ET, Kendzor DE. Mobile Health Interventions for Substance Use Disorders. Annu Rev Clin Psychol. 2024 Jul;20(1):49-76. doi: 10.1146/annurev-clinpsy-080822-042337. Epub 2024 Jul 2. PMID 38346293
- [Background] Businelle MS, Ma P, Kendzor DE, Frank SG, Vidrine DJ, Wetter DW. An Ecological Momentary Intervention for Smoking Cessation: Evaluation of Feasibility and Effectiveness. J Med Internet Res. 2016 Dec 12;18(12):e321. doi: 10.2196/jmir.6058. PMID 27956375
- [Background] Businelle MS, Lam CY, Kendzor DE, Cofta-Woerpel L, McClure JB, Cinciripini PM, Wetter DW. Alcohol consumption and urges to smoke among women during a smoking cessation attempt. Exp Clin Psychopharmacol. 2013 Feb;21(1):29-37. doi: 10.1037/a0031009. PMID 23379613
- [Background] Businelle MS, Kendzor DE, Reitzel LR, Costello TJ, Cofta-Woerpel L, Li Y, Mazas CA, Vidrine JI, Cinciripini PM, Greisinger AJ, Wetter DW. Mechanisms linking socioeconomic status to smoking cessation: a structural equation modeling approach. Health Psychol. 2010 May;29(3):262-73. doi: 10.1037/a0019285. PMID 20496980
- [Background] Bryant J, Bonevski B, Paul C, McElduff P, Attia J. A systematic review and meta-analysis of the effectiveness of behavioural smoking cessation interventions in selected disadvantaged groups. Addiction. 2011 Sep;106(9):1568-85. doi: 10.1111/j.1360-0443.2011.03467.x. Epub 2011 Jul 22. PMID 21489007
- [Background] Brandon TH, Vidrine JI, Litvin EB. Relapse and relapse prevention. Annu Rev Clin Psychol. 2007;3:257-84. doi: 10.1146/annurev.clinpsy.3.022806.091455. PMID 17716056
- [Background] Boland VC, Stockings EA, Mattick RP, McRobbie H, Brown J, Courtney RJ. The Methodological Quality and Effectiveness of Technology-Based Smoking Cessation Interventions for Disadvantaged Groups: A Systematic Review and Meta-analysis. Nicotine Tob Res. 2018 Feb 7;20(3):276-285. doi: 10.1093/ntr/ntw391. PMID 28034998
- [Background] Boland VC, Mattick RP, McRobbie H, Siahpush M, Courtney RJ. "I'm not strong enough; I'm not good enough. I can't do this, I'm failing"- A qualitative study of low-socioeconomic status smokers' experiences with accesssing cessation support and the role for alternative technology-based support. Int J Equity Health. 2017 Nov 13;16(1):196. doi: 10.1186/s12939-017-0689-5. PMID 29132364
- [Background] Bodin F, McIntyre KM, Schwartz JE, McKinley PS, Cardetti C, Shapiro PA, Gorenstein E, Sloan RP. The Association of Cigarette Smoking With High-Frequency Heart Rate Variability: An Ecological Momentary Assessment Study. Psychosom Med. 2017 Nov/Dec;79(9):1045-1050. doi: 10.1097/PSY.0000000000000507. PMID 28731984
- [Background] Bertz JW, Epstein DH, Preston KL. Combining ecological momentary assessment with objective, ambulatory measures of behavior and physiology in substance-use research. Addict Behav. 2018 Aug;83:5-17. doi: 10.1016/j.addbeh.2017.11.027. Epub 2017 Nov 16. PMID 29174666
- [Background] Benowitz NL, Bernert JT, Foulds J, Hecht SS, Jacob P, Jarvis MJ, Joseph A, Oncken C, Piper ME. Biochemical Verification of Tobacco Use and Abstinence: 2019 Update. Nicotine Tob Res. 2020 Jun 12;22(7):1086-1097. doi: 10.1093/ntr/ntz132. PMID 31570931
- [Background] Bell BM, Alam R, Alshurafa N, Thomaz E, Mondol AS, de la Haye K, Stankovic JA, Lach J, Spruijt-Metz D. Automatic, wearable-based, in-field eating detection approaches for public health research: a scoping review. NPJ Digit Med. 2020 Mar 13;3:38. doi: 10.1038/s41746-020-0246-2. eCollection 2020. PMID 32195373
- [Background] Battalio SL, Conroy DE, Dempsey W, Liao P, Menictas M, Murphy S, Nahum-Shani I, Qian T, Kumar S, Spring B. Sense2Stop: A micro-randomized trial using wearable sensors to optimize a just-in-time-adaptive stress management intervention for smoking relapse prevention. Contemp Clin Trials. 2021 Oct;109:106534. doi: 10.1016/j.cct.2021.106534. Epub 2021 Aug 8. PMID 34375749
- [Background] Alharbi R, Shahi S, Cruz S, Li L, Sen S, Pedram M, Romano C, Hester J, Katsaggelos AK, Alshurafa N. SmokeMon: Unobtrusive Extraction of Smoking Topography Using Wearable Energy-Efficient Thermal. Proc ACM Interact Mob Wearable Ubiquitous Technol. 2022 Dec;6(4):155. doi: 10.1145/3569460. Epub 2023 Jan 11. PMID 38031552
- [Background] Al-Khalidi FQ, Saatchi R, Burke D, Elphick H, Tan S. Respiration rate monitoring methods: a review. Pediatr Pulmonol. 2011 Jun;46(6):523-9. doi: 10.1002/ppul.21416. Epub 2011 Jan 31. PMID 21560260
- [Background] Adler NE, Newman K. Socioeconomic disparities in health: pathways and policies. Health Aff (Millwood). 2002 Mar-Apr;21(2):60-76. doi: 10.1377/hlthaff.21.2.60. PMID 11900187
- [Derived] El-Toukhy S, Haghayegh S, Leavens E, Sassano F, Tarran R. Use of non-invasive wearables biomonitoring to detect presmoking, smoking and postsmoking stages: protocol for an observational laboratory study. BMJ Open. 2025 Aug 16;15(8):e103292. doi: 10.1136/bmjopen-2025-103292. PMID 40819863